CLINICAL TRIAL: NCT02727361
Title: Role of the Striatal Cholinergic System in the Pathophysiology of Dystonia
Acronym: DYSCHOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX2014/20
Record Dates: First submitted 2016-03-21; First posted 2016-04-04 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Dystonia
Keywords: Dystonia; Binding potential; FEOBV
MeSH Terms: conditions — Dystonia | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cholinergic striatal imaging (Experimental): Cholinergic striatal imaging (IRM and TEP) to compare the intensity of the binding of cholinergic tracer
  Interventions: Radiation: PET (Positron Emission Tomography) imaging; Other: MRI : Magnetic Resonance Imaging

INTERVENTIONS:
Radiation: PET (Positron Emission Tomography) imaging — Molecular imaging using a PET radiotracer of the vesicular acetylcholine transporter.
Other: MRI : Magnetic Resonance Imaging — Multimodal MRI, MRI diffusion tensor (to study the microscopic structure of white matter) and functional MRI of the resting state (to study the functional organization of cerebral cholinergic networks at rest).

SUMMARY:
Dystonia is defined as a syndrome of sustained muscle contractions resulting in repetitive movements and abnormal postures. DYT1 is the most common form of genetic dystonia, but the link between genomic mutations and phenotypic expression remains largely unknown. Furthermore, secondary forms of dystonia have highlighted the role of the basal ganglia, particularly the putamen in the pathophysiology of the disease. Experimental results in a genetic model of dystonia in rodents suggest that cholinergic inter-neurons (ACh-I) of the putamen play a critical role in the pathological process of plasticity in the cortico-striatal synapse. However, these results have not been demonstrated in humans.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that the phenotype of dystonia is associated with the degree of striatal ACh-I alterations.

In this molecular imaging study, the investigators will directly test this hypothesis using a PET radiotracer of the vesicular acetylcholine transporter (VAT). Their goal is to explore the relationships between cholinergic dysfunction and clinical disease expression and the associated morphological and functional alterations. The experimental protocol will also include multimodal MRI, MRI diffusion tensor (to study the microscopic structure of white matter) and functional MRI of the resting state (to study the functional organization of cerebral cholinergic networks at rest).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 18 to 75 years, with health insurance European health insurance card (for resident patients in EU), insurance by bilateral social security agreement signed between his country and France (for resident patients outside the EU)
* Diagnosis of dystonia DYT1 confirmed by molecular biology (TORSINE- A gene mutation)
* Patient who stopped his anticholinergic treatment 48 hours before imaging

Exclusion Criteria:

* Patients who underwent surgery for deep brain stimulation or under cholinergic treatment.
* Presence of a counter-indication for MRI
* Presence of a counter-indication for TEP Scan with [18F]-FEOBV
* Woman premenopausal without effective ongoing contraception (intrauterine device or combined hormonal)
* Patient who underwent a PET examination in the previous month
* Presence of any health problem preventing travel to the imaging service of the University Hospital
* Being under the legal guardianship of another person or being unable to provide consent to participate
* Pregnant or breastfeeding woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Binding potential | Inclusion (V0)
  Image (PET) of the intensity of fixation of Cholinergic tracer (Binding potential)

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDEZ Philippe, Principal Investigator — University Hospital, Bordeaux; BURBAUD Pierre, Study Chair — University of Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France